CLINICAL TRIAL: NCT05202028
Title: Comparison of the Efficacy of Abdominal Massage, Connective Tissue Massage and Reflexology Applications on Constipation and Sleep Quality in Children With Cerebral Palsy
Brief Title: The Efficacy of Massage and Reflexology Applications in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Elif İrem Günaydın, PT, MSc, Halic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/015
Record Dates: First submitted 2022-01-08; First posted 2022-01-21 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy; Chronic Constipation
Keywords: Cerebral Palsy; Chronic constipation; sleep quality
MeSH Terms: conditions — Cerebral Palsy; Sleep Initiation and Maintenance Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Classic abdominal massge (Experimental): After the physical therapy applied to the patient by the physiotherapist in the special education center, 3 days a week for 8 weeks, once a day for approximately 15-20 minutes. Classic abdominal massage will be applied. To families; Training will be given on sleep hygiene, nutritional recommendations and lifestyle changes.
  Interventions: Other: Classic abdominal massage
- Connective tissue massage (Experimental): After the physical therapy applied to the patient by the physiotherapist in the special education center, 3 days a week for 8 weeks, once a day for approximately 15-20 minutes. Connective tissue massage will be applied. To families; Training will be given on sleep hygiene, nutritional recommendations and lifestyle changes.
  Interventions: Other: Connective Tissue Massage
- Reflexology (Experimental): After the physical therapy applied to the patient by the physiotherapist in the special education center for 8 weeks, 3 days a week for about 15-20 minutes. reflexology will be practiced. To families; Training will be given on sleep hygiene, nutritional recommendations and lifestyle changes.
  Interventions: Other: Reflexology

INTERVENTIONS:
Other: Reflexology — After the physical therapy applied to the patient by the physiotherapist in the special education center for 8 weeks, 3 days a week for about 15-20 minutes. reflexology will be practiced. To families; Training will be given on sleep hygiene, nutritional recommendations and lifestyle changes.
  Arms: Reflexology
Other: Connective Tissue Massage — After the physical therapy applied to the patient by the physiotherapist in the special education center, 3 days a week for 8 weeks, once a day for approximately 15-20 minutes. Connective tissue massage will be applied. To families; Training will be given on sleep hygiene, nutritional recommendations and lifestyle changes.
  Arms: Connective tissue massage
Other: Classic abdominal massage — After the physical therapy applied to the patient by the physiotherapist in the special education center for 8 weeks, 3 days a week for about 15-20 minutes. reflexology will be practiced. To families; Training will be given on sleep hygiene, nutritional recommendations and lifestyle changes.
  Arms: Classic abdominal massge

SUMMARY:
The study aims to compare the effectiveness of classical massage, connective tissue massage, and reflexology in children with cerebral palsy.

DETAILED DESCRIPTION:
The universe of the study will consist of children aged 4-18 years with a diagnosis of CP and chronic constipation who were admitted to the Duha Special Education and Rehabilitation Center. As a result of the power analysis, the minimum number of participants was determined as 20 for each group. Measurement and evaluation will be made to the groups three times, before the study, after the study (8th week), and follow-up at the 12th week.

Evaluations will be made by another physiotherapist who has no knowledge of the research topic and research groups. Children participating in the study will be determined by randomization using the closed-envelope method. The study is a randomized controlled experimental study.

In the study, the effects of treatments on the level of constipation, participation inactivity, and patient-parent sleep quality will be questioned. The sociodemographic data of the participants will be recorded in the general evaluation form. Gross Motor Function Classification System (KMFSS) to classify motor function levels, Gross Motor Function Scale-88 (KMFF-88) to assess functional status, and Functional Independence Measure= FIM to assess spasticity, Modified Ashworth Scale to assess constipation, Bristol for constipation assessment The Poo Scale and Constipation Severity Scale (BSS), and the Child Sleep Form (CUF) and the Pittsburgh Sleep Quality Index (PUKI) will be used for sleep assessment.

1. Group - Classical Abdominal Massage Group: After the physical therapy applied to the patient by the physiotherapist in the special education center, 3 days a week for 8 weeks, once a day for approximately 15-20 minutes. Classic abdominal massage will be applied. To families; Training will be given on sleep hygiene, nutritional recommendations, and lifestyle changes.
2. Group- Connective Tissue Massage Group: After the physical therapy applied to the patient by the physiotherapist in the special education center for 8 weeks, 3 days a week, once a day for approximately 15-20 minutes. Connective tissue massage will be applied. To families; Training will be given on sleep hygiene, nutritional recommendations, and lifestyle changes.
3. Group- Reflexology Group: After the physical therapy applied to the patient by the physiotherapist in the special education center for 8 weeks, 3 days a week for approximately 15-20 minutes. reflexology will be practiced. To families; Training will be given on sleep hygiene, nutritional recommendations, and lifestyle changes.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with cerebral palsy
* According to Gross Motor Function Test III, IV. and level V.
* Constipation in the last 6 months
* Age range is 4-18 years old
* Absence of any cardiopulmonary disease that will prevent exercise
* Patients who were informed about the study and whose families gave written consent to participate in the study will be included in the study.

Exclusion Criteria:

* Having undergone surgery involving intestinal health
* Having a chronic infectious bowel disease
* Having a congenital intestinal anomaly
* To have received Botox treatment in the last 6 months
* Absence of constipation in the last 6 months
* Levels I and II according to Gross Motor Function Test
* Having uncontrolled epileptic seizures
* Not signing the voluntary information and consent form
* Not continuing to work regularly

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Gross Motor Function Measure (GMFM-88) at 8 weeks and 12 weeks | At the beginning of study, 8th week of study and 12th week of study
  Gross Motor Function Scale-88 (GMFF-88) was created to evaluate changes in gross motor functions as growth and development continue in individuals with CP. It is a standardized, regular, systematic observational test. There are consecutive categories during normal motor and physiological development. These; supine, prone, crawling, sitting, laptop, standing, walking, and use of stairs. These categories include activities suitable for the titles in the sub-items. Scoring is divided into five main categories. It consists of a total of 88 items, 17 in the supine and prone categories, 20 in the sitting category, 14 in the crawling and kneeling category, 13 in the standing category, 24 in the walking-running and stair-climbing category. While testing these items, gross motor functions are correctly evaluated according to the level of achievement.
Change from Baseline in Functional Independence Measure (FIM) at 8 weeks and 12 weeks | At the beginning of study, 8th week of study and 12th week of study
  It is a method developed in 1993 by making use of the Functional Independence Measure (FIM) developed by the Uniform Data System for Medical Rehabilitation (UDS) system for adults. FIM; It is used in the entire adulthood, starting from the age of 10, after acquired events such as stroke, head trauma, spinal cord injury. WeeFIM was originally developed to evaluate the function of children aged 6 months to 7 years with congenital disorders. In a later study, it was proven that it is a valid and reliable method for children aged 6 months to 12 years, which can be used both in preschool and school age. Validity and reliability study in Turkey by Tur et al. made by. WeeFIM contains a total of 18 items in 6 areas: self-care, sphincter control, transfers, locomotion, communication, social and cognitive.
Change from Baseline in Bristolian Scale (BS) at 8 weeks and 12 weeks | At the beginning of study, 8th week of study and 12th week of study
  The Bristolian Scale is a 7-point scale used to describe stool consistency. He divides the stool structure into seven headings:
  1. Pieces like split hard nuts
  2. Sausage-shaped pieces with hard lumpy surface
  3. Pieces with cracks in the surface, such as sausages or snakes
  4. Soft pieces with smooth surface, such as sausages or snakes
  5. Pieces of fluffy feces with irregular sharp edges
  6. Flaky pieces with irregular edges
  7. Juicy, no solid parts The Bristolian Scale has been shown to be associated with colonic transit time in children with and without constipation. Hard stools fit 1 and 2, loose (ideal) stools fit 3, 4, 5, and diarrhea type 6 and 7. Therefore, it was represented as hard, loose stools and diarrhea according to stool consistency scores.
Change from Baseline in Constipation Severity Scale (CSS) at 8 weeks and 12 weeks | At the beginning of study, 8th week of study and 12th week of study
  Varma MG in 2008 to measure the severity of constipation. et al. Developed by The KCS is a scale that questions the frequency, intensity and strain of defecation in individuals. This scale, which can provide information about the symptoms of constipation, consists of 16 questions. Its Turkish validity and reliability were evaluated by Nurten Kaya et al. There are basically 3 sections in the survey conducted by Stool Obstruction, Large Intestine Laziness and Pain. BCS scores between 0 and 73, and high values indicate the severity of constipation.
Change from Baseline in Sleep Form in Children (SFC) at 8 weeks and 12 weeks | At the beginning of study, 8th week of study and 12th week of study
  This form, which was prepared to evaluate the sleep status of children, was prepared by Ronald Chervin et al. It was developed by Dr. to assess sleep-related problems in children aged 2-18 years. There is a short version of the scale consisting of 22 questions, as well as a long version consisting of 72 questions. Oner et al. There are three parts in the scale, the validity and reliability of which has been tested by (30). Part A (behaviors observed at night and during sleep time) consists of 43 questions, part B (behaviors observed during the day and possible problems) consists of 23 questions, and part C (attention deficit and hyperactivity) consists of 6 questions. Answers to the questions in sections A and B are given as 'yes', 'no' or 'I don't know'. The questions in section C are in 4-point Likert type. While scoring the C section, markings 0 and 1 are recoded as zero, markings 2 and 3 are recoded as one point. 22 items are used in scoring the scale.
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) at 8 weeks and 12 weeks | At the beginning of study, 8th week of study and 12th week of study
  PUKI, Buysse et al. It was developed by Ağargün et al. It was adapted into Turkish by in 1996. PUKI is a 19-item self-report scale that evaluates sleep quality and disturbance in the past month. It consists of 24 questions, 19 questions self-report questions, 5 questions to be answered by the spouse or roommate. The 18 scored questions of the scale consist of 7 components. Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disorder, Sleeping Drug Use, and Daytime Dysfunction. Each component is evaluated over 0-3 points. The total score of the 7 components gives the scale total score. The total score ranges from 0 to 21. A total score greater than 5 indicates "poor sleep quality".

SECONDARY OUTCOMES:
Change from Baseline in Modifiye Ashworth Scale (MAS) at 8 weeks and 12 weeks | At the beginning of study, 8th week of study and 12th week of study
  The Modified Ashworth Scale (MAS) is one of the most commonly used methods for measuring spasticity. The resistance to the movement made by moving the joint passively, rapidly and repetitively is scored. The MAS application is frequently used in studies because it is simple and can be practiced without the need for any tools. In MAS, it is a 6-point scale in which the patient grades resting muscle tone from the lowest grade "normal" to the highest grade "rigid" according to personal opinion.
  0: No increase in tone
  1. Slight increase in tone described by catching or minimal resistance at the end of NEH 1+: Mild increase in tone described with minimal resistance in less than half of the ROM
  2. Significant increase in tone but full range of motion in most ROMs
  3. Significant increase in muscle tone, difficulty in passive movement
  4. Joint is rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: Elif İrem Günaydın, PT, MSc, Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esmel-Esmel N, Tomas-Esmel E, Tous-Andreu M, Bove-Ribe A, Jimenez-Herrera M. Reflexology and polysomnography: Changes in cerebral wave activity induced by reflexology promote N1 and N2 sleep stages. Complement Ther Clin Pract. 2017 Aug;28:54-64. doi: 10.1016/j.ctcp.2017.05.003. Epub 2017 May 12. PMID 28779938
- [Background] Holey LA, Dixon J. Connective tissue manipulation: a review of theory and clinical evidence. J Bodyw Mov Ther. 2014 Jan;18(1):112-8. doi: 10.1016/j.jbmt.2013.08.003. Epub 2013 Sep 8. PMID 24411158